CLINICAL TRIAL: NCT03608917
Title: Efficacy and Safety of Total Glucosides of Paeony Combined With NB-UVB in the Treatment of Sporadic Vitiligo in Proceeding: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Total Glucosides of Paeony Combined With NB-UVB on Treating Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xjpfW (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); First Hospital of China Medical University (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, xjpfW, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XijingH-PF-20180116
Record Dates: First submitted 2018-07-04; First posted 2018-08-01 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Vitiligo
Keywords: Vitiligo; Total Glucosides of Paeony(TGP); narrow-band ultraviolet B (NB-UVB)
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Drug:Total Glucosides of Paeony (TGP)
  1. Time Frame: Week0-week8 The 1st Week, TGP 0.6g , Bid, orally; 2nd to Week8 , TGP 0.6g , Tid, orally combined with NB-UVB phototherapy( 1 time every other day)
  2. Time Frame: Week9-Week24 TGP, 0.6g, Tid, orally.
  Interventions: Drug: Total Glucosides of Paeony(TGP); Device: Narrow band-ultraviolet b（NB-UVB）
- Control group (Placebo Comparator): Drug:Total Glucosides of Paeony (TGP) analogue
  1. Time Frame:Week0-week8 The 1st Week, TGP analogue 0.6g , Bid, orally; 2nd to Week8, TGP analogue (0.6g , Tid, orally) combined with NB-UVB phototherapy( 1 time every other day)
  2. Time Frame: Week9-Week24 TGP analogue, 0.6g, Tid, orally.
  Interventions: Device: Narrow band-ultraviolet b（NB-UVB）; Drug: Total Glucosides of Paeony(TGP) analogue

INTERVENTIONS:
Drug: Total Glucosides of Paeony(TGP) — Total Glucosides of Paeony(TGP) as a traditional Chinese medicine, peony root is the dried root of peony of Ranunculaceae, cultivated all over the country.TGP is new drug of western medicine, original discovered by Professor Xu who is a famous pharmacologist. The main ingredient is a group of glycosides, including paeoniflorin, hydroxy paeoniflorin, paeoniflorin, paeoniflorin, benzoyl paeoniflorin etc, collectively referred to as total glucosides of paeony（TGP）
  Arms: Treatment group
Device: Narrow band-ultraviolet b（NB-UVB） — phototherapy on treating vitiligo
Drug: Total Glucosides of Paeony(TGP) analogue — Total Glucosides of Paeony(TGP) analogue as a placebo for Control group
  Arms: Control group

SUMMARY:
1. Total Glucosides of Paeony(TGP) As a traditional Chinese medicine, peony root is the dried root of peony of Ranunculaceae, cultivated all over the country.The main ingredient is a group of glycosides, including paeoniflorin, hydroxy paeoniflorin, paeoniflorin, paeoniflorin, benzoyl paeoniflorin etc, collectively referred to as total glucosides of paeony（TGP）. Paeoniflorin accounted for more than 90% of the TGP, is the main active ingredient of white peony root.By pharmacological and clinical studies of TGP, it have found that the mechanism of TGP is unique and mainly acts on the upstream of the immune response - inhibiting the presentation of antigens. It is different from immunosuppressive agents on T, B lymphocytes, or hormones and other drugs acting on the whole process.
2. Vitiligo Vitiligo is a pigment deprived skin disease caused by the destruction of melanocytes, the global incidence of about 1%. The pathogenesis is not yet clear, the current study shows that oxidative stress and autoimmunity is an important part of its occurrence and development.
3. The basic and clinical research of TGP used in vitiligo The ratio of cluster of differentiation 4+ / cluster designation 8+ T cell vs. cluster of differentiation 4+ chronotropic dose 25+ in the peripheral blood of patients with vitiligo could be significantly increase, after patients treatment by TGP combined with tacrolimus. Thereby enhancing the patient's maintenance of immune self-stability and Immune tolerance ability, promoting the healing of skin lesions. It showed significant effect in stable vitiligo,when patients treated by autologous epidermal grafting combined with TGP.

ELIGIBILITY:
Inclusion Criteria:

* subjects must be clinically diagnosed by the investigator to have sporadic Vitiligo in proceeding
* Vitiligo with at least 3 depigmented areas in different anatomy areas including：1%~50% of the total body surface area (BSA) in （face /trunk/limbs）,the minimum area is greater than 1 cm2 .Males or females, 18 Years to 65 Years of age at the time of signing the informed consent document.

.Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

* Actively spreading vitiligo,or stable vitiligo;
* Subjects with segmental, acromegaly, mucous, generalized, mixed and undetermined vitiligo.;
* Secondary vitiligo subjects with history of UV photosensitivity
* Subjects with other diseases unsuitable for ultraviolet light therapy and TGP ; .Use of vitiligo topical drugs within 2 weeks or, system treatment and phototherapy for the treatment of vitiligo within four weeks.
* History of allergy to any component of the total glucosides of paeony(TGP);
* Subjects with a history of chronic diarrhea or peptic ulcer within 1 year .Women who are pregnant or breast feeding,or preparing for pregnancy. .Subjects with serious medical diseases or history of mental system abnormal. .Use of any prior and concomitant therapy not listed above that may interfere with the objective of the study as per discretion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Vitiligo Area and Severity Index (VASI) | Change from Baseline VASI at 24 weeks
  The extent of residual depigmentation is expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. The VASI for each body part is the product of the palm unit and the degree of depigmentation of the unit.VASI=Σall body sites (hand units) × depigmentation

SECONDARY OUTCOMES:
The number of recovered vitiligo area | 8 weeks
  The number of recovered vitiligo area

CONTACTS AND LOCATIONS:
Overall Officials: Tianwen Gao, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No